CLINICAL TRIAL: NCT03055767
Title: Effectiveness of Onabotulinumtoxin A (Botox) in Pediatric Patients Experiencing Migraines: A Randomized Double Blinded Placebo Cross-over Study in the Pediatric Pain Population
Brief Title: Effectiveness of Onabotulinumtoxin A (Botox) in Pediatric Patients Experiencing Migraines: A Study in the Pediatric Pain Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Shalini Suresh Shah, Vice Chair, Pain Management, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20163108; UCIANES09 (Other: University of California, Irvine)
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Migraine Disorders; Headache, Migraine; Pediatrics
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OnabotulinumtoxinA/Saline Placebo (Other): The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  Interventions: Drug: OnabotulinumtoxinA; Other: Placebo (Saline)
- Saline Placebo/OnabotulinumtoxinA (Other): The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  Interventions: Drug: OnabotulinumtoxinA; Other: Placebo (Saline)

INTERVENTIONS:
Drug: OnabotulinumtoxinA — The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  Other Names: Botox
Other: Placebo (Saline) — The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.

SUMMARY:
The purpose of the research is to examine the outcomes of pediatric patients receiving Botulinum toxin type A (Botox ®) for the treatment of migraine. There is limited literature on the effectiveness of Botox ® in the treatment of chronic neurological pain in pediatric patients, specifically in the treatment of migraines.

DETAILED DESCRIPTION:
Medical Literature approximates one in three children will experience chronic headaches in their lifetime, which increases as children reach adolescence. Migraines make up nearly 60% of all visits to a pediatric headache specialist. Studies have demonstrated the negative impact of having childhood migraine on overall quality of life is similar to pediatric cancer, heart disease and rheumatic disease. As the frequency of migraine attacks increase, so does proportionally the child's disability in lost school time and family and social interactions, all of which may lead in turn to economic disability. Studies estimate the health care costs are 70% higher for a family with a migraine than a non-migraine affected family, and direct medical costs for children with migraine are reported to be similar to those for adults. A study published in JAMA 2003 found that health care costs, work-related disability for parents and lost educational opportunity for the child leads to an annual economic impact in the US of approximately $36 billion due to both direct medical costs and lost productivity into adulthood.

Onaboutlinum (BOTOX) is currently FDA approved as a very successful treatment to prevent migraines in adults, however not yet children. Current treatments for migraine in children appear to be insufficient. No trials currently exist in literature prospectively studying onabotulinumtoxinA for efficacy and/or safety for indication of pediatric migraine, although significant contributions have been made by retrospective case series over the last 10 years.

This research will be the first investigator-initiated study to study BOTOX (R) in children prospectively in a randomized controlled placebo, cross-over study. The overriding rationale is to demonstrate efficacy, tolerability and safety of onabotulinumtoxinA for pediatric migraine and thereby potentially hasten the lengthy process to evaluate BOTOX® for approval in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 - 17 years of age with a history of migraine meeting the criteria established in ICHD-II (2004), Section 1. Patients will provide at least 28-day baseline data in the form in the daily diary and must have at least 15 days of reported headache during this period, with at least 4 distinct episodes lasting at least 4 hours each.

Exclusion Criteria:

* Previous use of botulinum toxin of any serotype for any reason
* Pregnancy.
* Diagnosis of Myasthenia gravis, Eaton Lambert Syndrome, Amyotrophic Lateral Sclerosis
* Treatment of headache using acupuncture, transcutaneous electrical stimulation (TENS), cranial traction, dental splints, or injection of anesthetics/steroids within 4 weeks prior to the week of screening visit

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalini S Shah, MD, Principal Investigator — Assistant Clinical Professor
Locations (2):
- United States (2):
  - Gottschalk Medical Plaza, Irvine, California
  - UC Irvine Medical Center, Orange, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aurora SK, Winner P, Freeman MC, Spierings EL, Heiring JO, DeGryse RE, VanDenburgh AM, Nolan ME, Turkel CC. OnabotulinumtoxinA for treatment of chronic migraine: pooled analyses of the 56-week PREEMPT clinical program. Headache. 2011 Oct;51(9):1358-73. doi: 10.1111/j.1526-4610.2011.01990.x. Epub 2011 Aug 29. PMID 21883197
- [Background] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038
- [Background] Ahmed K, Oas KH, Mack KJ, Garza I. Experience with botulinum toxin type A in medically intractable pediatric chronic daily headache. Pediatr Neurol. 2010 Nov;43(5):316-9. doi: 10.1016/j.pediatrneurol.2010.06.001. PMID 20933173
- [Background] Bonfert M, Straube A, Schroeder AS, Reilich P, Ebinger F, Heinen F. Primary headache in children and adolescents: update on pharmacotherapy of migraine and tension-type headache. Neuropediatrics. 2013 Feb;44(1):3-19. doi: 10.1055/s-0032-1330856. Epub 2013 Jan 9. PMID 23303551
- [Background] Brodsky JR, Cusick BA, Zhou G. Evaluation and management of vestibular migraine in children: Experience from a pediatric vestibular clinic. Eur J Paediatr Neurol. 2016 Jan;20(1):85-92. doi: 10.1016/j.ejpn.2015.09.011. Epub 2015 Oct 22. PMID 26521123
- [Background] Chan VW, McCabe EJ, MacGregor DL. Botox treatment for migraine and chronic daily headache in adolescents. J Neurosci Nurs. 2009 Oct;41(5):235-43. doi: 10.1097/jnn.0b013e3181aaa98f. PMID 19835236
- [Background] Hermann C, Kim M, Blanchard EB. Behavioral and prophylactic pharmacological intervention studies of pediatric migraine: an exploratory meta-analysis. Pain. 1995 Mar;60(3):239-55. doi: 10.1016/0304-3959(94)00210-6. PMID 7596620
- [Background] Hershey AD, Powers SW, Coffey CS, Eklund DD, Chamberlin LA, Korbee LL; CHAMP Study Group. Childhood and Adolescent Migraine Prevention (CHAMP) study: a double-blinded, placebo-controlled, comparative effectiveness study of amitriptyline, topiramate, and placebo in the prevention of childhood and adolescent migraine. Headache. 2013 May;53(5):799-816. doi: 10.1111/head.12105. Epub 2013 Apr 17. PMID 23594025
- [Background] Jacobs H, Gladstein J. Pediatric headache: a clinical review. Headache. 2012 Feb;52(2):333-9. doi: 10.1111/j.1526-4610.2011.02086.x. Epub 2012 Jan 30. PMID 22288433
- [Background] Kabbouche M, O'Brien H, Hershey AD. OnabotulinumtoxinA in pediatric chronic daily headache. Curr Neurol Neurosci Rep. 2012 Apr;12(2):114-7. doi: 10.1007/s11910-012-0251-1. PMID 22274570
- [Background] Kacperski J, Hershey AD. Preventive drugs in childhood and adolescent migraine. Curr Pain Headache Rep. 2014 Jun;18(6):422. doi: 10.1007/s11916-014-0422-7. PMID 24760491
- [Background] Yonker M, Mangum T. Migraine management in children. Curr Neurol Neurosci Rep. 2015 May;15(5):20. doi: 10.1007/s11910-015-0540-6. PMID 25772998
- [Background] Tajti J, Szok D, Csati A, Vecsei L. Prophylactic Drug Treatment of Migraine in Children and Adolescents: An Update. Curr Pain Headache Rep. 2016 Jan;20(1):1. doi: 10.1007/s11916-015-0536-6. PMID 26695061
- [Derived] Shah S, Calderon MD, Crain N, Pham J, Rinehart J. Effectiveness of onabotulinumtoxinA (BOTOX) in pediatric patients experiencing migraines: a randomized, double-blinded, placebo-controlled crossover study in the pediatric pain population. Reg Anesth Pain Med. 2021 Jan;46(1):41-48. doi: 10.1136/rapm-2020-101605. Epub 2020 Oct 26. PMID 33106278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric subjects aged 8 to 17 were recruited during an enrollment window from March 1st, 2017 to November 30th, 2018 at the UCI Health Center for Pain and Wellness located at UCI Health's Gottschalk Medical Plaza.
Groups:
- Cross-over: OnabotulinumtoxinA, Then Saline Placebo: The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second. Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
- Cross-over: Saline Placebo, Then OnabotulinumtoxinA: The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
- Open Label Botox: Following unblinding, subject elected Botox treatment for 24 week open-label period where all subjects receive Botox treatment.
- Open Label Standard of Care: Following unblinding, subject elected to a 24-week return to conservative management per standard-of-care protocols.
Period: Double-Blind Period
Arm/Group | Cross-over: OnabotulinumtoxinA, Then Saline Placebo | Cross-over: Saline Placebo, Then OnabotulinumtoxinA | Open Label Botox | Open Label Standard of Care
Started | 9 | 6 | 0 | 0
Completed | 9 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Open-Label Period
Arm/Group | Cross-over: OnabotulinumtoxinA, Then Saline Placebo | Cross-over: Saline Placebo, Then OnabotulinumtoxinA | Open Label Botox | Open Label Standard of Care
Started | 0 | 0 | 11 | 4
Completed | 0 | 0 | 9 | 3
Not Completed | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 15 subjects randomized into the baseline, double-blind period (cross-over).
Groups:
- Cross-Over: OnabotulinumtoxinA, Then Saline Placebo: The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  OnabotulinumtoxinA: The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  Placebo (Saline): The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
- Cross-Over: Saline Placebo, Then OnabotulinumtoxinA: The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  OnabotulinumtoxinA: The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
  Placebo (Saline): The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
- Total: Total of all reporting groups
Arm/Group | Cross-Over: OnabotulinumtoxinA, Then Saline Placebo | Cross-Over: Saline Placebo, Then OnabotulinumtoxinA | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 6 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Migraines
Description: The frequency of migraines in days.
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Baseline Period | Control: 4-Week baseline period prior to injection procedures.
- Botox Period: 12-Week period where subject receives onabotulinumtoxinA
- Placebo Period: 12-week period where subject receives placebo injections.
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
days | 28 [20 to 28] | 20 [7 to 28] | 28 [23 to 28]
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.038, Wilcoxon signed-rank test

2. Primary Outcome: Intensity of Migraines
Description: Median intensity of migraines based on 0-10 Pain Numeric Rating Score (NRS). The higher the score, the more intense the pain.
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | 8 [7 to 10] | 5 [3 to 7] | 7 [5 to 9]
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.047, Wilcoxon signed-rank test)

3. Primary Outcome: Migraine Duration, in Hours
Description: Duration of migraines in hours.
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
hours | 24 [13 to 24] | 10 [2 to 24] | 24 [4 to 24]
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.148, Wilcoxon signed-rank test)

4. Primary Outcome: Pediatric Migraine Disability Score (PedMIDAS)
Description: Pediatric Migraine Disability Score consists of 6 questions: 3 addressing school attendance and functioning, and 3 evaluating participation in events outside of school. The questionnaire is based on the patient's recall of the previous 3 months.
  The questionnaire produces a raw score (0-10, 11-30, 31-50, >50) corresponding to a disability grade with increasing severity (little to non, mild, moderate, and severe) which was coded (1, 2, 3, and 4).
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
score on a scale | 4 [4 to 4] | 3 [2 to 4] | 4 [4 to 4]
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.047, Wilcoxon signed-rank test)

5. Secondary Outcome: Functionality Improvement
Description: Improvement of functionality as determined by their Pediatric Migraine Disability Score (PedMIDAS). The PedMIDAS consists of 6 questions: 3 addressing school attendance and functioning, and 3 evaluating participation in events outside of school. The questionnaire is based on the patient's recall of the previous 3 months.
  The questionnaire produces a raw score (0-10, 11-30, 31-50, >50) corresponding to a disability grade with increasing severity (little to non, mild, moderate, and severe) which was coded (1, 2, 3, and 4).
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Population: Baseline acted as control so no data for Functionality Improvement collected from participants at baseline.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15
score on a scale | 1 [0 to 1] | 0 [-1 to 0]
Statistical Analysis 1: Comparison: Botox Period vs Placebo Period; Test type: Superiority; p = 0.002, Wilcoxon signed-rank test)

6. Secondary Outcome: Difficulty Sleeping
Description: Subject reported having difficulty sleeping
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
Participants | 12 | 5 | 11
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.82, McNemar

7. Secondary Outcome: Hospital Admissions
Description: Admission to hospital
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
Participants | 8 | 0 | 2
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.006, McNemar

8. Secondary Outcome: Emergency Department (ED) Visits
Description: Subject visited an Emergency Department
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
Participants | 8 | 2 | 3
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.039, McNemar

9. Secondary Outcome: Home School
Description: Subject is home schooled full-time.
Time Frame: Baseline (4 weeks) and 12 weeks post, respective intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
Participants | 2 | 2 | 2
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.016, McNemar

10. Secondary Outcome: School Plan Enrollment
Description: Subject is enrolled in a school plan such as IEP, 504 plan, or similar modified school schedule.
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
Participants | 11 | 10 | 10
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.18, McNemar

11. Secondary Outcome: Duration of Benefit
Description: The duration of benefit in weeks
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Population: No data collected from participants at 4-week baseline in order to act as the control.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15
weeks | 4 [0 to 10] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Botox Period vs Placebo Period; Test type: Superiority; p < 0.001, Wilcoxon signed-rank test)

12. Secondary Outcome: Concomitant Headache Medications
Description: Number of concomitant headache medications taken
Time Frame: Baseline (4 weeks) and 12 weeks post each, respective intervention
Measure: Median (Inter-Quartile Range); unit: number taken
Arm/Group | Baseline Period | Control | Botox Period | Placebo Period
Number analyzed (Participants) | 15 | 15 | 15
number taken | 3 [1 to 4] | 1 [0 to 4] | 2 [1 to 5]
Statistical Analysis 1: Comparison: Baseline Period | Control vs Botox Period vs Placebo Period; Test type: Superiority; p = 0.64, Wilcoxon signed-rank test)

13. Other Pre Specified Outcome: Frequency of Migraines | Open-label Period
Description: The frequency of migraines during the open-label period (2 additional rounds of onabotulinumtoxinA) as compared to the cross-over period.
Time Frame: 24-48 weeks post-baseline period
Population: 15 subjects completed the cross-over period. Of those 15, 11 continued Botox (2 lost to follow-up), and 4 elected conservative management (1 discontinued intervention)
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Open-Label Period | Standard-of-Care: Subjects unblinded and elected to continue with standard care pain consultation (conservative management).
- Open-Label Period | Botox Continued: Subjects unblinded and elected to continue with 2 additional rounds of onabotulinumtoxinA.
Arm/Group | Open-Label Period | Standard-of-Care | Open-Label Period | Botox Continued
Number analyzed (Participants) | 4 | 11
days | 28 [21 to 28] | 20 [5 to 28]

14. Other Pre Specified Outcome: Intensity of Migraines | Open-Label Period
Description: Intensity of migraines during the the open-label period (2 additional rounds of onabotulinumtoxinA) as compared to the cross-over period.
  Intensity based on 0-10 Pain Numeric Rating Score (NRS). The higher the score, the more intense the pain.
Time Frame: 24-48 weeks post-baseline period
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Cross-Over Period: 24-week double-blind period where subjects were randomized into Group A (Botox cross-over to Placebo) or Group B (Placebo cross-over to Botox)
Arm/Group | Cross-Over Period | Open-Label Period | Botox Continued | Open-Label Period | Standard-of-Care
Number analyzed (Participants) | 15 | 11 | 4
units on a scale | 8 [7 to 10] | 5 [4 to 7] | 6 [5 to 8]

15. Other Pre Specified Outcome: Pediatric Migraine Disability Score (PedMIDAS) | Open-Label Period
Description: The PedMIDAS the open-label period (2 additional rounds of onabotulinumtoxinA) as compared to the cross-over period.
  The PedMIDAS consists of 6 questions: 3 addressing school attendance and functioning, and 3 evaluating participation in events outside of school. The questionnaire is based on the patient's recall of the previous 3 months.
  The questionnaire produces a raw score (0-10, 11-30, 31-50, >50) corresponding to a disability grade with increasing severity (little to non, mild, moderate, and severe) which was coded (1, 2, 3, and 4).
Time Frame: 24-48 weeks post-baseline period
Population: After the unblinding visit, 11 subjects elected to continue with the open-label period and were scheduled to receive two additional rounds of OBTA treatment (2 were lost to follow up). 4 subjects elected to receive standard of care (1 discontinued intervention).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cross-Over Period | Open-Label Period | Botox Continued | Open-Label Period | Standard-of-Care
Number analyzed (Participants) | 12 | 9 | 3
score on a scale | 4 [4 to 4] | 3 [2 to 4] | 4 [3 to 4]

16. Other Pre Specified Outcome: Duration of Migraine | Open-Label Period
Description: Duration of migraine in hours during the open-label period (2 additional rounds of onabotulinumtoxinA) as compared to the cross-over period.
Time Frame: 24-48 weeks post-baseline period
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cross-Over Period | Open-Label Period | Botox Continued | Open-Label Period | Standard-of-Care
Number analyzed (Participants) | 12 | 9 | 3
hours | 24 [13 to 24] | 6 [2 to 14] | 24 [24 to 24]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Cross-over: OnabotulinumtoxinA/Saline Placebo: The AB subject group will receive OnabotulinumtoxinA in the first treatment and saline placebo in the second. Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study.
  Randomization will be via selection of sealed envelope.
- Cross-over: Saline Placebo/OnabotulinumtoxinA: The BA subject group will receive saline and then Onabotulinumtoxin. A.Both groups will then receive OnabotulinumtoxinA in the last two treatments. There will be one treatment at the beginning of each 12 week block, meaning 4 treatments over the 48 week study period total. Progress check-ups will occur every 6 weeks during the study. Randomization will be via selection of sealed envelope.
- Off Label Botox:: Following unblinding, subject elected Botox treatment for 24 week open-label period where all subjects receive Botox treatment.
- Off Label Standard of Care:: Following unblinding, subject elected to a 24-week return to conservative management per standard-of-care protocols.
Arm/Group | Cross-over: OnabotulinumtoxinA/Saline Placebo | Cross-over: Saline Placebo/OnabotulinumtoxinA | Off Label Botox: | Off Label Standard of Care:
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/9 | 0/3

LIMITATIONS AND CAVEATS:
A lack of diversity in subject demographics and age. Didn't control for patients seeking alternative therapies during the study period, nor attempt to control concomitant medications.

Patients with comorbidities can have an impact on the treatment effect. PedMIDAS may not account for seasonal changes or patients with modified school schedules.

Continuation of baseline therapy is a confounding variable. Pain diary records required follow-up. Data collection relied in part on subject recall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03055767/Prot_SAP_000.pdf